CLINICAL TRIAL: NCT02926599
Title: High Fidelity Simulation Performance After a Potential Optimization Training for Anesthesiologist Resident: a Randomized Controlled Trial.
Brief Title: Potential Optimization Training in Simulation.
Acronym: TOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, MD, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TOPCLESS
Record Dates: First submitted 2016-09-30; First posted 2016-10-06 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: High Fidelity Simulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personal Optimization Training (Experimental): Personal Optimization Training such as positive reinforcement, personalized psycho-physiological relaxation and mental rehearsal (total 5 hours a few weeks before the simulation).
  Having 2 min to focus on techniques they were trained, after briefing of the scenario and before the start of the scenario.
  Interventions: Behavioral: Personal Optimization Training
- Control (No Intervention): No particular training.
  Screening of normal labs results during 2 min, after briefing of the scenario and before the start of the scenario.

INTERVENTIONS:
Behavioral: Personal Optimization Training
  Arms: Personal Optimization Training

SUMMARY:
Simulated environment allowed safe learning of critical events and knowledge of appropriate response and treatment. Anesthesiology resident education curriculum in Lyon plans several high fidelity simulation session with a large panel of critical events. Anticipation of critical events before they may occur and planification of team resources and priority in the treatment strategy may help to improve team performance during the scenario. The investigators' goal is to compare individual and team performances with or without an optimization personal potential training.

DETAILED DESCRIPTION:
The investigators aim to compare the individual and team performances for resident who were taught personal optimization skills (positive reinforcement, personalized psycho-physiological relaxation, mental rehearsal) and those who didn't.

The investigators are going to compare groups of anesthesiology residents going through same scenarios of simulated critical events in high fidelity simulation session. Scenarios will be recorded to be analyzed by 2 reviewers independently. A specific checklist of appropriate treatment and a non technical skill checklist will be use to cote team performance (OTTAWA and TEAM scales). Stress of the participants will be assessed by visual analogic scale of participants anxiety and stress. The two groups will be compare to see if improvement in team performance is associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology and Intensive care resident in the simulation education curriculum

Exclusion Criteria:

* Refusal to participate (written approval required)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Performance during simulation | day 1
  Performance will be assessed by the sum of 3 assessment: Ottawa non technical skill scale, team scanle and specific technical skill scale Total will be a number from 0 to 100.

SECONDARY OUTCOMES:
visual analogic scale of anxiety | day 1
  Visual analogic scales of anxiety
Visual analogic scales of confidence | day 1
  Visual analogic scales of confidence

OTHER OUTCOMES:
psychometric POMS scales | day 1
  psychometric POMS scales
psychometric STAI scales | day 1
  psychometric STAI scales

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques, Lehot, PHD, Study Chair — CLESS
Locations (1):
- CLESS, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided